# STATISTICAL ANALYSIS PLAN Protocol 1VIT13036

A Multi-center, Open-Label, Single Arm Study to Characterize the Pharmacokinetics and Pharmacodynamics Profile of Intravenous Ferric Carboxymaltose in Pediatric Subjects 1-17 years old with Iron Deficiency Anemia (IDA)

Prepared for:
Luitpold Pharmaceuticals, Inc.
Clinical Research and Development
800 Adams Avenue, Suite 100
Norristown, PA 19403
(610) 650-4200

Prepared by:
MedTrials, Inc.
1400 N. Providence Road
Building 1, Suite 212
Media, PA 19063

# **Document Version History:**

| Version | Date | Author | Comments |
|---|---|---|---|
| 1.0 | 6/8/15 | Michelle Secic | Original |
| 2.0 | 7/14/15 | Michelle Secic | Revisions based on initial review from Luitpold |
| 2.1 | 2/4/17 | Michelle Secic | Excluded summary of potentially clinically significant (PCS) Vital Signs |

# TABLE OF CONTENTS

| LIS | ST OF ABBREVIATIONS | 4 |
|---|---|---|
| 1. | INTRODUCTION | 5 |
| 2. | STUDY OBJECTIVES | 5 |
| 3. | STUDY DESIGN | 5 |
| 4. | PLANNED ANALYSES 4.1. Interim Analyses 4.2. Final Analysis 4.3. Populations | 8<br>8 |
| 5. | SAMPLE SIZE CONSIDERATIONS | 8 |
| 6. | REPORTING CONVENTIONS | 9 |
| 7. | STATISTICAL ANALYSES AND SUMMARIES 7.1. General Statistical Considerations 7.2. Baseline Definitions 7.3. Subject Disposition 7.4. Demographic Characteristics 7.5. Medical/Surgical History 7.6. Efficacy 7.7. Adverse Events 7.8. Laboratory Values 7.9. Vital Signs | |
| AP | PPENDIX A – TABLE SHELLS | 11 |
| AP | PPENDIX B – LISTING SHELLS | 11 |

# LIST OF ABBREVIATIONS

| AE | Adverse event |
|--------|----------------------------------------------|
| AUC | Area Under the Curve |
| BMI | Body Mass Index |
| DSMB | Data and Safety Monitoring Board |
| EDC | Electronic Data Capture |
| ESA | Erythropoiesis stimulating agent |
| FCM | Ferric Carboxymaltose |
| HBsAg | Hepatitis B antigen |
| HCV | Hepatitis C viral antibody |
| HIV | Human Immunodeficiency Virus |
| ID | Iron deficiency |
| IDA | Iron deficiency anemia |
| IV | Intravenous |
| IWR | Interactive Web Response |
| MedDRA | Medical Dictionary for Regulatory Activities |
| PCS | Potentially Clinically Significant |
| PD | Pharmacodynamics |
| PK | Pharmacokinetics |
| PT | Preferred Term |
| SAE | Serious Adverse Event |
| SAP | Statistical analysis plan |
| SOC | System Organ Class |
| TEAE | Treatment emergent adverse event |
| TSAT | Transferrin Saturation |

### 1. INTRODUCTION

Rapid growth, insufficient dietary intake, and limited absorption of dietary iron combine to place children at increased risk for iron deficiency. In addition, iron deficiency may contribute significantly to anemia due to malabsorption, gastrointestinal blood loss, or iatrogenically due to repeated blood samplings. As a result, iron deficiency anemia (IDA) remains the most common nutritional deficiency in children in the United States.

## 2. STUDY OBJECTIVES

The main objectives of this study are to characterize the pharmacokinetics and determine appropriate dosing and safety of Ferric Carboxymaltose for the pediatric population suffering from iron deficiency (ID) with anemia.

The pharmacokinetics component has its own separate statistical analysis plan (SAP). This SAP is intended to provide details on the dosing and safety components of the study, including the statistical methodology and associated tables and listings.

## 3. STUDY DESIGN

This is a phase II, open-label, non-randomized, multi-center, single arm study with two cohorts:

Cohort 1: 16 subjects will be treated with Ferric Carboxymaltose at 7.5 mg/kg with a maximum single dose of 750 mg, whichever is smaller.

Cohort 2 will initiate enrollment only after all subjects in Cohort 1 have completed 4 weeks of therapy and a Data and Safety Monitoring Board (DSMB) approves continuation.

Cohort 2: 16 subjects will be treated with Ferric Carboxymaltose at 15 mg/kg with a maximum single dose of 750 mg, whichever is smaller.

## 3.1. Inclusion/Exclusion Criteria

As per section 4.2.1 in the protocol, the following are the study inclusion and exclusion criteria.

#### Inclusion Criteria:

- Male or female subjects 1 to 17 years of age (6 to 17 years of age in Russia only) with assent to participation and his/her parent or guardian is willing and able to sign the informed consent approved by the Independent Review Board / Ethics Committee.
- Screening TSAT < 20%</li>
- Screening Hemoglobin < 11 g/dL</li>
- 4. For subjects who are receiving an erythropoietin stimulating agent (ESA): stable ESA therapy (+/- 20% of current dose) for > 8 weeks prior to the qualifying screening visit and no ESA dosing or product changes anticipated for the length of the trial

#### Exclusion Criteria:

- Known hypersensitivity reaction to any component of Ferric Carboxymaltose.
- Subject previously randomized and treated in this study or any other clinical study of Ferric Carboxymaltose (FCM or VIT-45).
- Body mass index (BMI) ≤ 5<sup>th</sup> percentile for age
- 4. Male or Female subject I year of age weighing < 12kg.
- History of acquired iron overload, hemochromatosis or other iron accumulation disorders.
- Chronic kidney disease subjects on hemodialysis.
- 7. Screening Ferritin level > 300ng/mL
- Subjects with significant severe diseases of the liver, hemopoietic system, cardiovascular system, psychiatric disorder or other conditions which on the opinion of the investigator may place a subject at added risk.
- Any active infection.
- Known positive hepatitis B antigen (HBsAg) or hepatitis C viral antibody (HCV) with evidence of active hepatitis.
- Known positive HIV-1/HIV-2 antibodies (anti-HIV).
- Anemia due to reasons other than iron deficiency (i.e. hemoglobinopathy).
   Subjects treated with vitamin B12 or folic acid deficiency are permitted.
- 13. Intravenous iron and /or blood transfusion in the 4 weeks prior to screening.
- Immunosuppressive therapy that may lead to anemia (i.e. cyclophosphamide, azathioprine, mycophenolate mofetil). Note steroid therapy is permitted.
- Administration and / or use of an investigational product (drug or device) within 30 days of screening.
- 16. Alcohol or drug abuse within the past six months.
- 17. Female subjects who are pregnant or lactating, or sexually active female who are of childbearing potential not willing to use an acceptable form of contraceptive precautions during the study.
- 18. Subject is unable to comply with study assessments.

#### 3.2. **Schedule of Visits**

Subjects will have a screening period, baseline visit, 24, 48 and 72 hours post dosing visits, and visits at day 14, 28 and 35. The schedule of visits is summarized below:

| Visit Day | Screening<br>Period<br>(Up to 14<br>Days) | Day<br>-1 | Day<br>0 | 24 and 48<br>hours<br>post<br>dosing | 72 hours<br>post<br>dosing | Day 14<br>(week 2) | Day 28<br>(week 4) | Day 35<br>(week 5) |
|---|---|---|---|---|---|---|---|---|
| Informed<br>Consent | Х | | | | | | | |
| Assess entry<br>criteria | Х | | Х | | | | | |
| EDC | X | | X | | | | | X |
| Medical History | Х | | X | | | | | |
| Physical Exam | | | Х | | | | | X |
| Vital Signs <sup>6</sup> | Х | | Х | | X | X | X | X |
| Height / Weight | | | Х | | | | | |
| PK/PD Samples | | $X^2$ | $X^3$ | X <sup>4</sup> | X <sup>4</sup> | | | |
| Hematology,<br>Chemistry and<br>Iron Indices | х | | | | х | х | х | Х |
| Serum<br>pregnancy test | Х | | | | | | | |
| Concomitant<br>Medications | Х | | Х | | Х | Х | Х | Х |
| ESA Stability | х | | Х | | Х | X | X | X |
| Adverse Event<br>Assessments <sup>5</sup> | | | Х | Х | Х | Х | X | Х |
| Ferric<br>Carboxymaltose | | | Х | | | | | |

<sup>&</sup>lt;sup>1</sup> Includes clinical assessment of skin, cardiovascular, pulmonary, abdominal, and central nervous system

<sup>&</sup>lt;sup>2</sup> Blood samples drawn at 8am, 12pm and 8pm for subject iron profile

<sup>&</sup>lt;sup>3</sup> Blood samples PK/PD should be taken prior to Ferric Carboxymaltose dosing and additional samples for PK/PD should be taken at 1, 2, 6 and 12 hours post dosing.

Blood samples should be taken approximately the same time of day as the Day 0 samples were drawn

<sup>&</sup>lt;sup>5</sup> Adverse event assessments starting at the time of Ferric Carboxymaltose dosing

<sup>&</sup>lt;sup>6</sup> Sitting vital signs including blood pressure and heart rate should be collected immediately pre-dosing, immediately and 30 minutes post dosing. Body temperature will also be collected pre-dose only. Vital signs on non-dosing days include sitting heart rate and blood pressure only.

### 4. PLANNED ANALYSES

# 4.1. Interim Analyses

An interim analysis of the safety data is planned after the first cohort of 16 patients have completed through week 4 of the study. The purpose of the interim analysis is for the DSMB to review the interim data and to make recommendations to Luitpold Pharmaceuticals concerning the merits of continuing the study and the safety of continuing enrollment into cohort 2.

Refer to the DSMB Charter to details on the planned review of the interim data.

# 4.2. Final Analysis

The final planned data analyses will be performed after all subjects have completed the study and after the database is locked.

# 4.3. Populations

There will be two analysis populations:

- The Safety Population: The safety population includes all subjects who receive Ferric Carboxymaltose.
- The Pharmacokinetics and Pharmacodynamics (PK/PD) Population: The PK/PD population includes all subjects in the safety population who have evaluable iron profiles and no protocol violation that could affect the PK/PD of Ferric Carboxymaltose.

All summaries will be presented for the safety population. Only demographic characteristics will be summarized for the PK/PD population.

## 5. SAMPLE SIZE CONSIDERATIONS

Determination of sample size for this study was a compromise between obtaining sufficiently precise estimates of pharmacokinetic parameters and the ethics of including a large number of pediatric patients in an experiment. The precision of estimation can be quantified as the width of the 95% confidence interval for area under the curve (AUC) from 0 to 72 (AUC $_{0-72}$ ) from this single-arm study (i.e., smaller width indicates better precision). Based on Study VIT-IV-CL-002 in adults, the standard deviation for total serum iron AUC $_{0-72}$  following a 500 mg intravenous dose is approximately 300 mg-hour/mL. The width of a 95% confidence interval, using a standard deviation of 300 mg-hour/mL, is presented below for selected sample sizes.

As seen in the figure below, 16 patients appears to be a reasonable compromise between precision and number of exposed pediatric patients. Therefore, 32 subjects will be enrolled, with 16 subjects in each cohort. Within each cohort of 16 subjects there will be 8 subjects 1 to 6 years of age and 8 subjects >6 to 17 years of age. Subject enrollment and ages will be tracked and monitored via interactive web response (IWR) system.



## 6. REPORTING CONVENTIONS

Unless otherwise specified, standard descriptive statistics will be computed for measurements presented in summary tables. The standard descriptive statistics for continuous variables include: number of observations analyzed, mean, standard deviation, median, and range (minimum, and maximum). The standard descriptive statistics for categorical variables include: frequency distribution with the number and percent of subjects included in each category.

Calculation of percentage will use the denominator of the total number of subjects with non-missing data in the particular group of analysis population used in the data display unless otherwise specified.

All data listings, summaries, and statistical analyses will be generated using SAS® Version 9.1 or higher (SAS is registered trademarks of the SAS Institute Inc., Cary, NC, USA.)

# 7. STATISTICAL ANALYSES AND SUMMARIES

## 7.1. General Statistical Considerations

No formal hypothesis testing is planned for this study. Only descriptive, summary statistics are planned for assessment of dosing and safety.

## 7.2. Baseline Definitions

Baseline for this study is defined as Day 0. If the data is not captured at Day 0, or if the data at Day 0 is missing, the screening value will be used.

# 7.3. Subject Disposition

Subject disposition will be summarized as: enrolled/registered, treated, completed or discontinued. For those discontinued, the reason for discontinuation will be summarized.

# 7.4. Demographic Characteristics

Demographic characteristics will be summarized separately for the treatment groups, and separately for the two study populations (safety and PK/PD). Demographic characteristics will include: age, gender, ethnicity and race.

# 7.5. Medical/Surgical History

Medical/surgical histories will be summarized separately for the treatment groups. System organ class and condition/surgery will be coded with the Medical Dictionary for Regulatory Activities (MedDRA) Terminology.

# 7.6. Efficacy

Hemoglobin, ferritin and TSAT will be summarized at each visit, and for each treatment group. In addition, the change from baseline to each visit will be summarized for each treatment group.

## 7.7. Adverse Events

Adverse events (AEs) will be summarized for treatment emergent adverse events (TEAEs). TEAEs are defined as AEs that occur on or after the day of the first dose. MedDRA terminology will be used to classify all AEs with respect to system organ class (SOC) and preferred term (PT).

A summary of subjects with TEAEs will be presented for each treatment group. The summary will include counts and percentages for subjects who experience at least one AE, overall and by SOC and PT. This will be repeated for severe TEAEs, related TEAEs and serious TEAEs. Severity will be captured as Grade 1 through Grade 5 with Grades 3-5 categorized as severe. Related will be captured as: none, unlikely, possibly or probably, with related = possibly or probably. Serious will be captured with the standard serious adverse event (SAE) criteria.

Subjects who report the same PT on multiple occasions will be counted once for the preferred term under the highest severity when summarizing by severity, under the closest relationship to the drug when summarizing by relationship, under most serious when summarizing by seriousness.

# 7.8. Laboratory Values

Laboratory values will be summarized at each visit, and for each treatment group. In addition, the change from baseline to each visit, and the incidence of treatment-emergent potentially clinically significant (PCS) laboratory values will be summarized for each treatment group.

## 7.9. Vital Signs

Vital signs will be summarized at each visit, and for each treatment group and by age groups (1 - < 6 years, and 6-17 years). Height and weight will be summarized at Day 0 only. Blood pressure and heart rate will be summarized at all visits and as the change from pre to immediately post treatment and the change from pre to 30 minutes post-treatment.

## APPENDIX A - TABLE SHELLS

```
Table 14.1.1 Site and Population Summaries

Table 14.1.1 Subject Disposition – Safety Population

Table 14.1.2.1 Demographic Characteristics – Safety Population

Table 14.1.2.2 Demographic Characteristics – PK/PD Population

Table 14.1.3 Medical/Surgical History – Safety Population

Table 14.2.1 Efficacy – Safety Population

Table 14.2.2 Summary of Intolerance and ESA – Safety Population

Table 14.3.1.1 Summary of Subjects with TEAEs – Safety Population

Table 14.3.1.2 Occurrence of TEAEs – Safety Population

Table 14.3.1.3 Occurrence of Severe TEAEs – Safety Population

Table 14.3.1.4 Occurrence of Related TEAEs – Safety Population

Table 14.3.1.5 Occurrence of Serious TEAEs – Safety Population

Table 14.3.2.1 Laboratory Values – Safety Population

Table 14.3.2.2 Incidence of Potentially Clinically Significant (PCS) Laboratory Values

Table 14.3.3.1 Vital Signs – Safety Population
```

## APPENDIX B-LISTING SHELLS

```
Listing 16.2.1.1 Completion/Discontinuation
Listing 16.2.1.2 Identification of Subjects with Clinically Important Protocol Violations
Listing 16.2.1.3 Inclusion/Exclusion Criteria
Listing 16.2.1.4 Patient Populations
Listing 16.2.1.5 Demographics
Listing 16.2.1.6 Medical/Surgical History
Listing 16.2.1.7 Drug Allergy/Intolerance at Screening
Listing 16.2.1.8 IV Iron Intolerance
Listing 16.2.1.9 Physical Examination
Listing 16.2.1.10 Iron Deficiency
Listing 16.2.2.1 Erythropoiesis Stimulating Agent
Listing 16.2.2.2 Ferric Carboxymaltoses Administration
Listing 16.2.2.3 Pharmacokinetic Samples
Listing 16.2.3.1 Concomitant Medications
Listing 16.2.3.2.1 Central Laboratory Values - CFR
Listing 16.2.3.2.2 Central Laboratory Values – Lab Transfer
```

Listing 16.2.3.2.3 Potentially Clinically Significant Central Laboratory Values - Lab Transfer

Listing 16.2.3.3.1 Vital Signs

Listing 16.2.3.4 Adverse Event Details

# STATISTICAL ANALYSIS PLAN Protocol 1VIT13036

A Multi-center, Open-Label, Single Arm Study to Characterize the Pharmacokinetics and Pharmacodynamics Profile of Intravenous Ferric Carboxymaltose in Pediatric Subjects 1-17 years old with Iron Deficiency Anemia (IDA)

Prepared for:
Luitpold Pharmaceuticals, Inc.
Clinical Research and Development
800 Adams Avenue, Suite 100
Norristown, PA 19403
(610) 650-4200

Prepared by:
MedTrials, Inc.
1400 N. Providence Road
Building 1, Suite 212
Media, PA 19063

# **Document Version History:**

| Version | Date | Author | Comments |
|---|---|---|---|
| 1.0 | 6/8/15 | Michelle Secic | Original |
| 2.0 | 7/14/15 | Michelle Secic | Revisions based on initial review from Luitpold |
| 2.1 | 6/17/16 | Michelle Secic | Revised to exclude PCS vitals and stratify by age instead |
| 2.2 | 6/21/16 | Michelle Secic | Revised section 7.9 as per Luitpold comments |
| 2.3 | 6/23/16 | Michelle Secic | Revised sections 7.5 and 7.8 as per Luitpold |
| 2.4 | 6/23/16 | Michelle Secic | Revised vital signs table to include additional changes over time |
| 2.5 | 6/24/16 | Michelle Secic | Split vital signs table |
| FINAL | 7/7/16 | Michelle Secic | Finalized date and version |

# TABLE OF CONTENTS

| LIS | ST OF A | ABBREVIATIONS | 4 |
|---|---|---|---|
| 1. | INTR | ODUCTION | 5 |
| 2. | STUD | OY OBJECTIVES | 5 |
| 3. | STUD<br>3.1.<br>3.2. | OY DESIGN Inclusion/Exclusion Criteria Schedule of Visits | 5 |
| 4. | PLAN<br>4.1.<br>4.2.<br>4.3. | INED ANALYSESInterim AnalysesFinal AnalysisPopulations | 8 |
| 5. | SAMI | PLE SIZE CONSIDERATIONS | 8 |
| 6. | REPO | RTING CONVENTIONS | 9 |
| 7. | STAT 7.1. 7.2. 7.3. 7.4. 7.5. 7.6. 7.7. 7.8. 7.9. | ISTICAL ANALYSES AND SUMMARIES General Statistical Considerations Baseline Definitions Subject Disposition Demographic Characteristics Medical/Surgical History Efficacy Adverse Events Laboratory Values Vital Signs | 9<br>10<br>10<br>10<br>10 |
| AP. | PENDI | X A – TABLE SHELLS | 2 |
| ΑP | PENDI | X B – LISTING SHELLS | 2 |

# LIST OF ABBREVIATIONS

| AE | Adverse event |
|--------|----------------------------------------------|
| AUC | Area Under the Curve |
| BMI | Body Mass Index |
| DSMB | Data and Safety Monitoring Board |
| EDC | Electronic Data Capture |
| ESA | Erythropoiesis stimulating agent |
| FCM | Ferric Carboxymaltose |
| HBsAg | Hepatitis B antigen |
| HCV | Hepatitis C viral antibody |
| HIV | Human Immunodeficiency Virus |
| ID | Iron deficiency |
| IDA | Iron deficiency anemia |
| IV | Intravenous |
| IWR | Interactive Web Response |
| MedDRA | Medical Dictionary for Regulatory Activities |
| PCS | Potentially Clinically Significant |
| PD | Pharmacodynamics |
| PK | Pharmacokinetics |
| PT | Preferred Term |
| SAE | Serious Adverse Event |
| SAP | Statistical analysis plan |
| SOC | System Organ Class |
| TEAE | Treatment emergent adverse event |
| TSAT | Transferrin Saturation |

## 1. INTRODUCTION

Rapid growth, insufficient dietary intake, and limited absorption of dietary iron combine to place children at increased risk for iron deficiency. In addition, iron deficiency may contribute significantly to anemia due to malabsorption, gastrointestinal blood loss, or iatrogenically due to repeated blood samplings. As a result, iron deficiency anemia (IDA) remains the most common nutritional deficiency in children in the United States.

## 2. STUDY OBJECTIVES

The main objectives of this study are to characterize the pharmacokinetics and determine appropriate dosing and safety of Ferric Carboxymaltose for the pediatric population suffering from iron deficiency (ID) with anemia.

The pharmacokinetics component has its own separate statistical analysis plan (SAP). This SAP is intended to provide details on the dosing and safety components of the study, including the statistical methodology and associated tables and listings.

## 3. STUDY DESIGN

This is a phase II, open-label, non-randomized, multi-center, single arm study with two cohorts:

Cohort 1: 16 subjects will be treated with Ferric Carboxymaltose at 7.5 mg/kg with a maximum single dose of 750 mg, whichever is smaller.

Cohort 2 will initiate enrollment only after all subjects in Cohort 1 have completed 4 weeks of therapy and a Data and Safety Monitoring Board (DSMB) approves continuation.

Cohort 2: 16 subjects will be treated with Ferric Carboxymaltose at 15 mg/kg with a maximum single dose of 750 mg, whichever is smaller.

## 3.1. Inclusion/Exclusion Criteria

As per section 4.2.1 in the protocol, the following are the study inclusion and exclusion criteria.

#### Inclusion Criteria:

- Male or female subjects 1 to 17 years of age (6 to 17 years of age in Russia only)
  with assent to participation and his/her parent or guardian is willing and able to
  sign the informed consent approved by the Independent Review Board / Ethics
  Committee.
- 2. Screening TSAT < 20%
- 3. Screening Hemoglobin < 11 g/dL
- 4. For subjects who are receiving an erythropoietin stimulating agent (ESA): stable ESA therapy (+/- 20% of current desc) for > 8 weeks prior to the qualifying screening visit and no ESA dosing or product changes anticipated for the length of the trial

### Exclusion Criteria:

- 1. Known hypersensitivity reaction to any component of Ferric Carboxymaltose,
- Subject previously randomized and treated in this study or any other clinical study of Ferric Carboxymaltose (FCM or VIT-45).
- 3. Body mass index (BMI)  $\leq 5^{m}$  percentile for age
- 4. Male or Female subject 1 year of age weighing < 12kg.
- Flistory of acquired iron overload, hemochromatosis or other iron accumulation disorders.
- 6. Chronic kidney disease subjects on hemodialysis.
- 7. Screening Ferritin level > 300ng/mL
- Subjects with significant severe diseases of the liver, hemopoietic system, cardiovascular system, psychiatric disorder or other conditions which on the opinion of the investigator may place a subject at added risk.
- 9. Any active infection.
- Known positive hepatitis B antigen (HBsAg) or hepatitis C viral antibody (HCV) with evidence of active hepatitis.
- 11. Known positive HIV-1/HIV-2 antibodies (anti-HIV),
- Anemia due to reasons other than iron deficiency (i.e. homoglobinopathy).
   Subjects treated with vitamin B12 or folic acid deficiency are permitted.
- 13. Intravenous iron and /or blood transfusion in the 4 weeks prior to screening.
- Immunosuppressive therapy that may lead to anemia (i.e. cyclophosphamide, azathioprine, mycophenolate mofetil). Note steroid therapy is permitted.
- Administration and for use of an investigational product (drug or device) within 30 days of screening.
- 16. Alcohol or drug abuse within the past six months.
- 17. Female subjects who are pregnant or lactating, or sexually active female who are of childbearing potential not willing to use an acceptable form of contraceptive precautions during the study.
- 18. Subject is unable to comply with study assessments.

# 3.2. Schedule of Visits

Subjects will have a screening period, baseline visit, 24, 48 and 72 hours post dosing visits, and visits at day 14, 28 and 35. The schedule of visits is summarized below:

| Visit Day | Screening Period (Up to 14 Days) | Day<br>-1 | Day<br>0 | 24 and 48<br>hours<br>post<br>dosing | 72 hours<br>post<br>dosing | Day 14<br>(week 2) | Day 28<br>(week 4) | Day 35 (week 5) |
|---|---|---|---|---|---|---|---|---|
| Informed<br>Consent | Х | | | | | | | |
| Assess entry criteria | Х | | Х | | | | | |
| EDC | Х | | Х | | | | | Х |
| Medical History | Х | | Х | | | | | |
| Physical Exam | | | X | | | | | Х |
| Vital Signs <sup>6</sup> | Х | | Х | | Х | X | X | Х |
| Height / Weight | | | X | | | | | |
| PK/PD Samples | | X3 | X <sup>s</sup> | X4 | X* | | | |
| Hematology,<br>Chemistry and<br>Iron Indices | Х | | | | Х | Х | Х | Х |
| Serum<br>pregnancy test | Х | | | | | | | |
| Concomitant<br>Medications | Х | | Х | | Х | Х | Х | Х |
| ESA Stability | Х | | Х | | Х | X | X | Х |
| Adverse Event Assessments <sup>3</sup> | | | Х | Х | х | X | Χ | Х |
| Ferric<br>Carboxymaltose | | | х | | | | | |

<sup>1</sup> Includes clinical assessment of skin, cardiovascular, pulmonary, abdominal, and central nervous system

<sup>2</sup>Blood samples drawn at 8am, 12pm and 8pm for subject iron profile

5 Adverse event assessments starting at the time of Ferric Carboxymaltose dosing

<sup>&</sup>lt;sup>3</sup> Blood samples PK/PD should be taken prior to Ferric Carboxymaltose dosing and additional samples for PK/PD should be taken at 1, 2, 6 and 12 hours post dosing.

Blood samples should be taken approximately the same time of day as the Day 0 samples were drawn

<sup>&</sup>lt;sup>6</sup> Sitting vital signs including blood pressure and heart rate should be collected immediately pre-dosing, immediately and 30 minutes post dosing. Body temperature will also be collected pre-dose only. Vital signs on non-dosing days include sitting heart rate and blood pressure only.

## 4. PLANNED ANALYSES

# 4.1. Interim Analyses

An interim analysis of the safety data is planned after the first cohort of 16 patients have completed through week 4 of the study. The purpose of the interim analysis is for the DSMB to review the interim data and to make recommendations to Luitpold Pharmaceuticals concerning the merits of continuing the study and the safety of continuing enrollment into cohort 2.

Refer to the DSMB Charter to details on the planned review of the interim data.

# 4.2. Final Analysis

The final planned data analyses will be performed after all subjects have completed the study and after the database is locked.

# 4.3. Populations

There will be two analysis populations:

- The Safety Population: The safety population includes all subjects who receive Ferric Carboxymaltose.
- The Pharmacokinetics and Pharmacodynamics (PK/PD) Population: The PK/PD population includes all subjects in the safety population who have evaluable iron profiles and no protocol violation that could affect the PK/PD of Ferric Carboxymaltose.

All summaries will be presented for the safety population. Only demographic characteristics will be summarized for the PK/PD population.

# 5. SAMPLE SIZE CONSIDERATIONS

Determination of sample size for this study was a compromise between obtaining sufficiently precise estimates of pharmacokinetic parameters and the ethics of including a large number of pediatric patients in an experiment. The precision of estimation can be quantified as the width of the 95% confidence interval for area under the curve (AUC) from 0 to 72 (AUC<sub>0-72</sub>) from this single-arm study (i.e., smaller width indicates better precision). Based on Study VIT-IV-CL-002 in adults, the standard deviation for total serum iron AUC<sub>0-72</sub> following a 500 mg intravenous dose is approximately 300 mg-hour/mL. The width of a 95% confidence interval, using a standard deviation of 300 mg-hour/mL, is presented below for selected sample sizes.

As seen in the figure below, 16 patients appears to be a reasonable compromise between precision and number of exposed pediatric patients. Therefore, 32 subjects will be enrolled, with 16 subjects in each cohort. Within each cohort of 16 subjects there will be 8 subjects 1 to 6 years of age and 8 subjects >6 to 17 years of age. Subject enrollment and ages will be tracked and monitored via interactive web response (IWR) system.



## 6. REPORTING CONVENTIONS

Unless otherwise specified, standard descriptive statistics will be computed for measurements presented in summary tables. The standard descriptive statistics for continuous variables include: number of observations analyzed, mean, standard deviation, median, and range (minimum, and maximum). The standard descriptive statistics for categorical variables include: frequency distribution with the number and percent of subjects included in each category.

Calculation of percentage will use the denominator of the total number of subjects with non-missing data in the particular group of analysis population used in the data display unless otherwise specified.

All data listings, summaries, and statistical analyses will be generated using SAS® Version 9.1 or higher (SAS is registered trademarks of the SAS Institute Inc., Cary, NC, USA.)

## 7. STATISTICAL ANALYSES AND SUMMARIES

# 7.1. General Statistical Considerations

No formal hypothesis testing is planned for this study. Only descriptive, summary statistics are planned for assessment of dosing and safety.

## 7.2. Baseline Definitions

Baseline for this study is defined as Day 0. If the data is not captured at Day 0, or if the data at Day 0 is missing, the screening value will be used.

# 7.3. Subject Disposition

Subject disposition will be summarized as: enrolled/registered, treated, completed or discontinued. For those discontinued, the reason for discontinuation will be summarized.

# 7.4. Demographic Characteristics

Demographic characteristics will be summarized separately for the treatment groups, and separately for the two study populations (safety and PK/PD). Demographic characteristics will include: age, gender, ethnicity and race.

# 7.5. Medical/Surgical History

Medical/surgical histories will be summarized separately for the treatment groups. System organ class and condition/surgery will be coded with the Medical Dictionary for Regulatory Activities (MedDRA) Terminology.

# 7.6. Efficacy

Hemoglobin, ferritin and TSAT will be summarized at each visit, and for each treatment group. In addition, the change from baseline to each visit will be summarized for each treatment group.

## 7.7. Adverse Events

Adverse events (AEs) will be summarized for treatment emergent adverse events (TEAEs). TEAEs are defined as AEs that occur on or after the day of the first dose. MedDRA terminology will be used to classify all AEs with respect to system organ class (SOC) and preferred term (PT).

A summary of subjects with TEAEs will be presented for each treatment group. The summary will include counts and percentages for subjects who experience at least one AE, overall and by SOC and PT. This will be repeated for severe TEAEs, related TEAEs and serious TEAEs. Severity will be captured as Grade 1 through Grade 5 with Grades 3-5 categorized as severe. Related will be captured as: none, unlikely, possibly or probably, with related = possibly or probably. Serious will be captured with the standard serious adverse event (SAE) criteria.

Subjects who report the same PT on multiple occasions will be counted once for the preferred term under the highest severity when summarizing by severity, under the closest relationship to the drug when summarizing by relationship, under most serious when summarizing by seriousness.

# 7.8. Laboratory Values

Laboratory values will be summarized at each visit, and for each treatment group. In addition, the change from baseline to each visit, and the incidence of treatment-emergent potentially clinically significant (PCS) laboratory values will be summarized for each treatment group. The denominator is all subjects with normal baseline (< Grade III value) and at least one post baseline assessment in the safety population and the numerator is the number of subjects with

PCS (i.e., meets Grade III or Grade IV toxicity criteria from the National Cancer Institute Common Terminology Criteria) at post-baseline.

# 7.9. Vital Signs

Vital signs will be summarized for dosing day (Day 0), at each visit and for each treatment group. The change from baseline to each visit, will be summarized for each treatment group. In addition, summary statistics for vital signs will be stratified by age groups: 1 - <6 years, and 6 to 17 years.

## APPENDIX A – TABLE SHELLS

- Table 14.1.1 Site and Population Summaries
- Table 14.1.1 Subject Disposition Safety Population
- Table 14.1.2.1 Demographic Characteristics Safety Population
- Table 14.1.2.2 Demographic Characteristics PK/PD Population
- Table 14.1.3 Medical/Surgical History Safety Population
- Table 14.2.1 Efficacy Safety Population
- Table 14.2.2 Summary of Intolerance and ESA Safety Population
- Table 14.3.1.1 Summary of Subjects with TEAEs Safety Population
- Table 14.3.1.2 Occurrence of TEAEs Safety Population
- Table 14.3.1.3 Occurrence of Severe TEAEs Safety Population
- Table 14.3.1.4 Occurrence of Related TEAEs Safety Population
- Table 14.3.1.5 Occurrence of Serious TEAEs Safety Population
- Table 14.3.2.1 Laboratory Values Safety Population
- Table 14.3.2.2 Incidence of Potentially Clinically Significant (PCS) Laboratory Values
- Table 14.3.3.1 Vital Signs Day 0 Safety Population
- Table 14.3.3.2 Vital Signs All Visits Safety Population

## APPENDIX B - LISTING SHELLS

- Listing 16.2.1.1 Completion/Discontinuation
- Listing 16.2.1.2 Identification of Subjects with Clinically Important Protocol Violations
- Listing 16.2.1.3 Inclusion/Exclusion Criteria
- Listing 16.2.1.4 Patient Populations
- Listing 16.2.1.5 Demographics
- Listing 16.2.1.6 Medical/Surgical History
- Listing 16.2.1.7 Drug Allergy/Intolerance at Screening
- Listing 16.2.1.8 IV Iron Intolerance
- Listing 16.2.1.9 Physical Examination
- Listing 16.2.1.10 Iron Deficiency
- Listing 16.2.2.1 Erythropoiesis Stimulating Agent
- Listing 16.2.2.2 Ferric Carboxymaltose Administration
- Listing 16.2.2.3 Pharmacokinetic Samples
- Listing 16.2.3.1 Concomitant Medications
- Listing 16.2.3.2.1 Central Laboratory Values CFR
- Listing 16.2.3.2.2 Central Laboratory Values Lab Transfer
- Listing 16.2.3.2.3 Potentially Clinically Significant Central Laboratory Values Lab Transfer
- Listing 16.2.3.3.1 Vital Signs
- Listing 16.2.3.4 Adverse Event Details

Luitpold Pharmaceuticals, Inc. SAP Version FINAL Protocol 1VIT13036

## Appendix A - Shells for Study Tables

## **Table of Contents**

| Table 14.1.1 Site and Population Summaries | 2 |
|---|---|
| Table 14.1.1 Subject Disposition – Safety Population | 3 |
| Table 14.1.2.1 Demographic Characteristics – Safety Population | 4 |
| Table 14.1.2.2 Demographic Characteristics – PK/PD Population | 5 |
| Table 14.1.3 Medical/Surgical History – Safety Population | 6 |
| Table 14.2.1 Efficacy – Safety Population | 7 |
| Table 14.2.2 Summary of Intolerance and ESA – Safety Population | 10 |
| Table 14.3.1.1 Summary of Subjects with TEAEs – Safety Population | 11 |
| Table 14.3.1.2 Occurrence of TEAEs – Safety Population | 12 |
| Table 14.3.1.3 Occurrence of Severe TEAEs – Safety Population | 13 |
| Table 14.3.1.4 Occurrence of Related TEAEs – Safety Population | 14 |
| Table 14.3.1.5 Occurrence of Serious TEAEs – Safety Population | 15 |
| Table 14.3.2.1 Laboratory Values – Safety Population | 16 |
| Table 14.3.2.2 Incidence of Potentially Clinically Significant (PCS) Laboratory Values | 18 |
| Table 14.3.3.1 Vital Signs – Day 0 – Safety Population | 20 |
| Table 14.3.3.2 Vital Signs – All Visits – Safety Population | 21 |


Table 14.1.1 Site and Population Summaries

| | Cohort 1 | Cohort 2 |
|----------------------|----------|----------|
| Site | X | X |
| Site #1 | X | X |
| Site #2 | X | X |
| Etc. | X | X |
| In Safety Population | X | Х |
| In PK Population | X | X |


Table 14.1.1 Subject Disposition - Safety Population

| | Cohort 1 | Cohort 2<br>(N=XXX) |
|-----------------------------|----------|---------------------|
| Disposition | (N=XXX) | |
| Registered/Enrolled | X (XX.X) | X (XX.X) |
| Completed Study | X (XX.X) | X (XX.X) |
| Discontinued due to: | X (XX.X) | X (XX.X) |
| Adverse Event | X (XX.X) | X (XX.X) |
| Intervention | X (XX.X) | X (XX.X) |
| Lost to Follow-up | X (XX.X) | X (XX.X) |
| Physician Decision | X (XX.X) | X (XX.X) |
| Withdrawal by Subject | X (XX.X) | X (XX.X) |
| Death | X (XX.X) | X (XX.X) |
| Study Terminated by Sponsor | X (XX.X) | X (XX.X) |
| Other | X (XX.X) | X(XX.X) |


Luitpold Pharmaceuticals, Inc. SAP Version FINAL Protocol 1VIT13036

Table 14.1.2.1 Demographic Characteristics – Safety Population

| Baseline Characteristic | Statistic | Cohort 1<br>(N=XXX) | Cohort 2<br>(N=XXX) |
|---|---|---|---|
| Age | N | XX | XX |
| Ago | Mean (SD) | XX (XX.X) | XX (XX.X) |
| | Median | XX | XX |
| | Range | XX, XX | XX, XX |
| Gender | Male | X (XX.X) | X (XX.X) |
| | Female | X (XX.X) | X (XX.X) |
| Ethnicity | Hispanic or Latino | X (XX.X) | X (XX.X) |
| | Not Hispanic or Latino | X (XX.X) | X (XX.X) |
| Race [1] | American Indian/Alaska Native | X (XX.X) | X (XX.X) |
| | Asian | X (XX.X) | X (XX.X) |
| | Black/African American | X (XX.X) | X (XX.X) |
| | Native Hawaiian/Other Pacific Islander | X (XX.X) | X (XX.X) |
| | White | X (XX.X) | X (XX.X) |

<sup>[1]</sup> Total may be more than 100% as this category is "check all that apply."


Luitpold Pharmaceuticals, Inc. SAP Version FINAL Protocol 1VIT13036

Table 14.1.2.2 Demographic Characteristics – PK/PD Population

| | | Cohort 1 | Cohort 2 |
|---|---|---|---|
| Baseline Characteristic | Statistic | (N=XXX) | (N=XXX) |
| Age | N | XX | XX |
| | Mean (SD) | XX (XX.X) | XX (XX.X) |
| | Median | XX | XX |
| | Range | XX, XX | XX, XX |
| Gender | Male | X (XX.X) | X (XX.X) |
| | Female | X (XX.X) | X (XX.X) |
| Ethnicity | Hispanic or Latino | X (XX.X) | X (XX.X) |
| | Not Hispanic or Latino | X (XX.X) | X (XX.X) |
| Race [1] | American Indian/Alaska Native | X (XX.X) | X (XX.X) |
| | Asian | X (XX.X) | X (XX.X) |
| | Black/African American | X (XX.X) | X (XX.X) |
| | Native Hawaiian/Other Pacific Islander | X (XX.X) | X (XX.X) |
| | White | X (XX.X) | X (XX.X) |

<sup>[1]</sup> Total may be more than 100% as this category is "check all that apply."


Table 14.1.3 Medical/Surgical History - Safety Population

| | | Cohort 1 | Cohort 2 |
|-----------------------|----------------------|----------|----------|
| System Organ Class | Condition/Surgery | (N=XXX) | (N=XXX) |
| System Organ Class #1 | Condition/Surgery #1 | X (XX.X) | X (XX.X) |
| | Condition/Surgery#2 | X(XX.X) | X (XX.X) |
| | Etc. | | |
| System Organ Class #2 | Condition/Surgery #1 | X (XX.X) | X(XX.X) |
| | Condition/Surgery #2 | X (XX.X) | X(XX.X) |
| | Etc. | | |
| Etc. | Condition/Surgery #1 | X (XX.X) | X(XX,X) |
| | Condition/Surgery #2 | X(XXX) | X(XX.X) |
| | Etc. | | |

Table 14.2.1 Efficacy - Safety Population

| Parameter | Visit | Statistic[1] | Cohort 1 (N=XXX) | Cohort 2<br>(N=XXX) |
|---|---|---|---|---|
| Hemoglobin | Screening | N | XX | XX |
| J | | Mean (SD) | XX (XX.X) | XX (XX.X) |
| | | Median | XX | XX |
| | | Range | XX, XX | XX, XX |
| | 72 hours post-dose | N | XX | XX |
| | 72 Hours post dose | Mean (SD) | XX (XX.X) | XX (XX.X) |
| | | Median | XX | XX |
| | | Range | XX, XX | XX, XX |
| | Change from Screening to 72 hours post-dose | N | XX | XX |
| | Change from Screening to 72 hours post-dose | Mean (SD) | XX (XX.X) | |
| | | Median | XX | XX (XX.X) |
| | | | | XX |
| | 5 44 | Range | XX, XX | XX, XX |
| | Day 14 | N | XX | XX |
| | | Mean (SD) | XX (XX.X) | XX (XX.X) |
| | | Median | XX | XX |
| | | Range | XX, XX | XX, XX |
| | Change from Screening to Day 14 | N | XX | XX |
| | | Mean (SD) | XX (XX.X) | XX (XX.X) |
| | | Median | XX | XX |
| | | Range | XX, XX | XX, XX |
| | Day 28 | N | XX | XX |
| | • | Mean (SD) | XX (XX.X) | XX (XX.X) |
| | | Median | XX | XX |
| | | Range | XX, XX | XX, XX |
| | Change from Screening to Day 28 | N | XX | XX |
| | enange nom eereening to 2 ay 20 | Mean (SD) | XX (XX.X) | XX (XX.X) |
| | | Median | XX | XX |
| | | Range | XX, XX | XX, XX |
| | Day 35 | N | XX | XX |
| | Day 33 | Mean (SD) | XX (XX.X) | XX (XX.X) |
| | | Median | XX | XX (XX.X) |
| | OL 6 0 : 1 D 25 | Range | XX, XX | XX, XX |
| | Change from Screening to Day 35 | N<br>N | XX | XX |
| | | Mean (SD) | XX (XX.X) | XX (XX.X) |
| | | Median | XX | XX |
| | | Range | XX, XX | XX, XX |
| erritin | Screening | Ν | XX | XX |
| | | Mean (SD) | XX (XX.X) | XX (XX.X) |
| | | Median | XX | XX |
| | | Range | XX, XX | XX, XX |
| | 72 hours post-dose | N | XX | XX |
| | | Mean (SD) | XX (XX.X) | XX (XX.X) |
| | | Median | XX | ХХ |
| | | Range | XX, XX | XX, XX |
| | Change from Screening to 72 hours post-dose | N | XX | XX |
| | change from cereening to 12 hours post dose | Mean (SD) | XX (XX.X) | XX (XX.X) |
| | | 1.16011 (07) | (******) | (******) |
| | | Median | XX | XX |


Table 14.2.1 Efficacy – Safety Population

| | | Statistic[1] | (N=XXX) | (N=XXX) |
|---|---|---|---|---|
| | Day 14 | N | XX | XX |
| | | Mean (SD) | XX (XX.X) | XX (XX.X) |
| | | Median | XX | XX |
| | | Range | XX, XX | XX, XX |
| | Change from Screening to Day 14 | N | XX | XX |
| | | Mean (SD) | XX (XX.X) | XX (XX.X |
| | | Median | XX | XX |
| | | Range | XX, XX | XX, XX |
| | Day 28 | N | XX | XX |
| | Duj 20 | Mean (SD) | XX (XX.X) | XX (XX.X) |
| | | Median | XX | XX |
| | | Range | XX, XX | XX, XX |
| | Change from Savening to Day 29 | | | |
| | Change from Screening to Day 28 | N<br>Marin (SD) | XX | XX |
| | | Mean (SD) | XX (XX.X) | XX (XX.X) |
| | | Median | XX | XX |
| | | Range | XX, XX | XX, XX |
| | Day 35 | N | XX | XX |
| | | Mean (SD) | XX (XX.X) | XX (XX.X) |
| | | Median | XX | XX |
| | | Range | XX, XX | XX, XX |
| | Change from Screening to Day 35 | N | XX | XX |
| | | Mean (SD) | XX (XX.X) | XX (XX X) |
| | | Median | XX | XX |
| | | Range | XX, XX | XX, XX |
| ΓSAT | Screening | N | XX | XX |
| | | Mean (SD) | XX (XX.X) | XX (XX.X) |
| | | Median | XX | XX |
| | | Range | XX, XX | XX, XX |
| | 72 hours post-dose | N | XX | XX |
| | | Mean (SD) | XX (XX.X) | XX (XX.X) |
| | | Median | XX | XX |
| | | Range | XX, XX | XX, XX |
| | Change from Screening to 72 hours post-dose | N | XX | XX |
| | Change from Screening to 72 hours post-dose | Mean (SD) | XX (XX.X) | XX (XX.X) |
| | | Median | XX (XX.X) | XX |
| | | Range | XX, XX | XX, XX |
| | D 14 | - | | |
| | Day 14 | N (GD) | XX | XX |
| | | Mean (SD) | XX (XX.X) | XX (XX.X) |
| | | Median | XX | XX |
| | | Range | XX, XX | XX, XX |
| | Change from Screening to Day 14 | N | XX | XX |
| | | Mean (SD) | XX (XX.X) | XX (XX,X) |
| | | Median | XX | XX |
| | | Range | XX, XX | XX, XX |
| | Day 28 | N | XX | XX |
| | | Mean (SD) | XX (XX.X) | XX (XX.X) |
| | | Median | XX | XX |
| | | Range | XX, XX | XX, XX |
| | Change from Screening to Day 28 | N | XX | XX |
| | change from consening to Day 20 | Mean (SD) | XX (XX.X) | XX (XX.X) |
| | | Median | XX | XX |
| | | Range | XX, XX | XX, XX |

Table 14.2.1 Efficacy – Safety Population

| Parameter | Visit | Statistic[1] | Cohort 1<br>(N=XXX) | Cohort 2<br>(N=XXX) |
|---|---|---|---|---|
| | Day 35 | N | XX | XX |
| | Day 33 | Mean (SD) | XX (XX.X) | XX (XX.X) |
| | | Median | XX | XX |
| | | Range | XX, XX | XX, XX |
| | Change from Screening to Day 35 | N | XX | XX |
| | | Mean (SD) | XX (XX.X) | XX (XX.X) |
| | | Median | XX | XX |
| | | Range | XX, XX | XX, XX |


Luitpold Pharmaceuticals, Inc. SAP Version FINAL Protocol I VIT13036

Table 14.2.2 Summary of Intolerance and ESA – Safety Population

| | Cohort 1 | Cohort 2 |
|--------------------------|----------|----------|
| | (N=XXX) | (N=XXX) |
| Drug Allergy Intolerance | X (XX.X) | X (XX.X) |
| IV Iron Intolerance | X (XX.X) | X (XX.X) |
| ESA | X (XX.X) | X (XX.X) |
| ESA | Λ (ΛΛ.Λ) | |


Luitpold Pharmaceuticals, Inc. SAP Version FINAL Protocol 1VIT13036

Table 14.3.1.1 Summary of Subjects with TEAEs - Safety Population

| | Cohort 1<br>(N=XXX) | Cohort 2<br>(N=XXX) |
|---|---|---|
| Any Treatment-Emergent Adverse Event [1] | X (XX.X) | X (XX.X) |
| Serious | X(XX.X) | X (XX.X) |
| Severe [2] | X(XX,X) | X(XX,X) |
| Related to Study Drug [3] | X(XX,X) | X(XX.X) |

<sup>[1]</sup> If a subject experiences the same event more than once, the first occurrence is tabulated [2] Refers to CTCAE grade 3, 4, or 5.
[3] Related includes Possibly or Probably related to study drug.


Table 14.3.1.2 Occurrence of TEAEs - Safety Population

| MedDRA System Organ Class | MedDRA Preferred Term | Cohort 1<br>(N=XXX) | Cohort 2<br>(N=XXX) |
|---|---|---|---|
| SOC #1 | Any | X (XX.X) | X (XX.X) |
| | PT#I | X (XX.X) | X (XX.X) |
| | PT #2 | X(XX.X) | X (XX.X) |
| | PT #3 | X (XX.X) | X (XX.X) |
| | Etc. | | |
| SOC #2 | Any | X (XX.X) | X (XX.X) |
| | PT #1 | X (XX.X) | X (XX.X) |
| | PT #2 | X (XX.X) | X (XX.X) |
| | PT #3 | X(XX.X) | X (XX.X) |
| | Etc. | | |
| Etc. | | | |

All AEs in this table are treatment-emergent. The denominator for the calculation of the percentage is the number of subjects in the group and the numerator is the number of subjects in the group with at least one TEAE in the given system organ class or with the given preferred term. If a subject experiences the same event more than once, the first occurrence is tabulated.


Table 14.3.1.3 Occurrence of Severe TEAEs – Safety Population

| MedDRA System Organ Class | MedDRA Preferred Term | Cohort 1<br>(N=XXX) | Cohort 2<br>(N=XXX) |
|---|---|---|---|
| SOC #1 | Any | X (XX.X) | X (XX.X) |
| | PT #1 | X (XX.X) | X (XX.X) |
| | PT #2 | X (XX.X) | X (XX.X) |
| | PT #3 | X (XX.X) | X (XX.X) |
| | Etc. | | |
| SOC #2 | Any | X (XX.X) | X (XX.X) |
| | PT #1 | X (XX.X) | X (XX.X) |
| | PT #2 | X (XX.X) | X (XX.X) |
| | PT #3 | X (XX.X) | X (XX.X) |
| | Etc. | | |
| Etc. | | | |

All AEs in this table are severe (Grade 3, 4 or 5) and treatment-emergent. The denominator for the calculation of the percentage is the number of subjects in the group and the numerator is the number of subjects in the group with at least one TEAE in the given system organ class or with the given preferred term. If a subject experiences the same event more than once, the first occurrence is tabulated.


Table 14.3.1.4 Occurrence of Related TEAEs - Safety Population

| | | Cohort 1 | Cohort 2 |
|---------------------------|-----------------------|----------|----------|
| MedDRA System Organ Class | MedDRA Preferred Term | (N=XXX) | (N=XXX) |
| SOC #1 | Any | X (XX.X) | X (XX.X) |
| | PT #1 | X (XX.X) | X (XX.X) |
| | PT #2 | X (XX.X) | X (XX.X) |
| | PT #3 | X (XX.X) | X (XX.X) |
| | Etc. | | |
| SOC #2 | Any | X(XX.X) | X(XX.X) |
| | PT #1 | X (XX.X) | X (XX.X) |
| | PT #2 | X (XX.X) | X (XX.X) |
| | PT #3 | X (XX.X) | X (XX.X) |
| | Etc. | | |
| Etc. | | | |

All AEs in this table are related (possibly or probably) to study drug and treatment-emergent. The denominator for the calculation of the percentage is the number of subjects in the group and the numerator is the number of subjects in the group with at least one TEAE in the given system organ class or with the given preferred term. If a subject experiences the same event more than once, the first occurrence is tabulated.


Table 14.3.1.5 Occurrence of Serious TEAEs – Safety Population

| | | Cohort 1 | Cohort 2 |
|---------------------------|-----------------------|----------|----------|
| MedDRA System Organ Class | MedDRA Preferred Term | (N=XXX) | (N=XXX) |
| SOC #1 | Any | X (XX.X) | X (XX.X) |
| | PT #1 | X (XX.X) | X (XX.X) |
| | PT #2 | X (XX.X) | X (XX.X) |
| | PT #3 | X (XX.X) | X (XX.X) |
| | Etc. | | |
| SOC #2 | Any | X (XX.X) | X (XX.X) |
| | PT #1 | X (XX.X) | X (XX.X) |
| | PT #2 | X (XX.X) | X (XX.X) |
| | PT #3 | X (XX.X) | X (XX.X) |
| | Etc. | | _ |
| Etc | | | |

All AEs in this table are serious and treatment-emergent. The denominator for the calculation of the percentage is the number of subjects in the group and the numerator is the number of subjects in the group with at least one TEAE in the given system organ class or with the given preferred term. If a subject experiences the same event more than once, the first occurrence is tabulated.


Table 14.3.2.1 Laboratory Values - Safety Population

| Parameter | Visit | Statistic[1] | Cohort 1<br>(N=XXX) | Cohort 2<br>(N=XXX) |
|---|---|---|---|---|
| ab #1 | Screening | N | XX | XX |
| | | Mean (SD) | XX (XX.X) | XX (XX.X) |
| | | Median | XX | XX |
| | | Range | XX, XX | XX, XX |
| | 72 hours post-dose | N | XX | XX |
| | | Mean (SD) | XX (XX.X) | XX (XX.X) |
| | | Median | XX | XX |
| | | Range | XX, XX | XX, XX |
| | Change from Screening to 72 | N | XX | XX |
| | hours post-dose | Mean (SD) | XX (XX.X) | XX (XX.X) |
| | - ' - | Median | XX | XX |
| | | Range | XX, XX | XX, XX |
| | Day 14 | N | XX | XX |
| | Day 14 | Mean (SD) | XX (XX.X) | XX (XX.X) |
| | | Median | XX | XX |
| | | Range | XX, XX | XX, XX |
| | Change from Screening to Day | N | XX | XX |
| | 14 | Mean (SD) | XX (XX.X) | XX (XX.X) |
| | 1.7 | Median | XX | XX |
| | | Range | XX, XX | XX, XX |
| | Day 29 | N | XX | XX, XX |
| | Day 28 | Mean (SD) | XX (XX.X) | XX (XX.X) |
| | | Median | XX | XX |
| | Character Carrelland A. Davi | Range | XX, XX | XX, XX |
| | Change from Screening to Day | N<br>Marin (SD) | XX | XX |
| | 28 | Mean (SD) | XX (XX.X) | XX (XX.X) |
| | | Median | XX | XX |
| | | Range | XX, XX | XX, XX |
| | Day 35 | N | XX | XX |
| | | Mean (SD) | XX (XX.X) | XX (XX.X) |
| | | Median | XX | XX |
| | | Range | XX, XX | XX, XX |
| | Change from Screening to Day | N | XX | XX |
| | 35 | Mean (SD) | XX (XX.X) | XX (XX.X) |
| | | Median | XX | XX |
| | | Range | XX, XX | XX, XX |
| ab #2 | Screening | N | XX | XX |
| | | Mean (SD) | XX (XX.X) | XX (XX.X) |
| | | Median | XX | XX |
| | | Range | XX, XX | XX, XX |
| | 72 hours post-dose | N | XX | XX |
| | | Mean (SD) | XX (XX.X) | XX (XX.X) |
| | | Median | XX | XX |
| | | Range | XX, XX | XX, XX |
| | Change from Screening to 72 | N | XX | XX |
| | hours post-dose | Mean (SD) | XX (XX.X) | XX (XX.X) |
| | - | Median | XX | XX |
| | | Range | XX, XX | XX, XX |

Table 14.3.2.1 Laboratory Values - Safety Population

| Parameter | Visit | Statistic[t] | Cohort 1<br>(N=XXX) | Cohort 2<br>(N=XXX) |
|---|---|---|---|---|
| | Day 14 | N<br>Mean (SD)<br>Median | XX<br>XX (XX.X)<br>XX | XX<br>XX (XX.X)<br>XX |
| | Change from Screening to Day | Range<br>N | XX, XX<br>XX | XX, XX<br>XX |
| | 14 | Mean (SD)<br>Median<br>Range | XX (XX.X)<br>XX<br>XX, XX | XX (XX.X)<br>XX<br>XX, XX |
| | Day 28 | N<br>Mean (SD)<br>Median<br>Range | XX<br>XX (XX.X)<br>XX<br>XX, XX | XX<br>XX (XX.X)<br>XX<br>XX, XX |
| | Change from Screening to Day 28 | N<br>Mean (SD)<br>Median<br>Range | XX<br>XX (XX.X)<br>XX<br>XX, XX | XX<br>XX (XX.X)<br>XX<br>XX, XX |
| | Day 35 | N<br>Mean (SD)<br>Median<br>Range | XX<br>XX (XX.X)<br>XX<br>XX, XX | XX<br>XX (XX.X)<br>XX<br>XX, XX |
| | Change from Screening to Day 35 | N<br>Mean (SD)<br>Median<br>Range | XX<br>XX (XX.X)<br>XX<br>XX, XX | XX<br>XX (XX.X)<br>XX<br>XX, XX |
| Etc. | Etc. | N<br>Mean (SD)<br>Median<br>Range | XX<br>XX (XX.X)<br>XX<br>XX, XX | XX<br>XX (XX.X)<br>XX<br>XX, XX |


Table 14.3.2.2 Incidence of Potentially Clinically Significant (PCS) Laboratory Values

| | | Cohort 1 | Cohort 2 |
|-------------------|-----|----------|----------|
| Lab Test/Category | PCS | (N=XXX) | (N=XXX) |
| Lab #1 | No | X (XX.X) | X (XX.X) |
| | Yes | X (XX.X) | X(XX.X) |
| Lab #2 | No | X (XX.X) | X (XX.X) |
| | Yes | X(XX,X) | X(XX.X) |
| Etc. | | | |





Table 14.3.3.1 Vital Signs - Day 0 - Safety Population

| All Subjects Sitting Diastolic BP (mmHg) Day 0 Pre-Treatment N XX Mean (SD) XX (XX.X) Median XX Range XXX, XX Day 0 Immediately Post-Treatment N XX Mean (SD) XX (XX.X) Median XX Mean (SD) XX (XX.X) Median XX Range XX, XX | (n=XXX) |
|---|---|
| Day 0 Immediately Post-Treatment N XX Mean (SD) XX (XX.X) Median XX | XX |
| Day 0 Immediately Post-Treatment N XX Mean (SD) XX (XX.X) Median XX | XX (XX.X) |
| Day 0 Immediately Post-Treatment N XX Mean (SD) XX (XX.X) Median XX | XX |
| Mean (SD) XX (XX.X)<br>Median XX | XX, XX |
| Median XX | XX |
| | XX (XX.X) |
| Pange YY YY | XX |
| Range AA, AA | XX, XX |
| Change from Pre-Treatment to N XX Immediately Post-Treatment | XX |
| Mean (SD) XX (XX.X) | XX (XX.X) |
| Median XX | XX |
| Range XX, XX | XX, XX |
| Day 0 30 Minutes Post-Treatment N XX | xx |
| Mean (SD) XX (XX.X) | XX (XX.X) |
| Median XX | XX |
| Range XX, XX | XX, XX |
| Change from Pre-Treatment to 30 N XX Minutes Post-Treatment | XX |
| Mean (SD) XX (XX.X) | XX (XX.X) |
| Median XX | XX |
| Range XX, XX | XX, XX |

Note to programmer, repeat above for all Systolic BP and Heart Rate and for two age stratum: 1 - < 6 years, and 6 - 17 years

Table 14.3.3.2 Vital Signs – All Visits – Safety Population

| Age Group | Vital Sign | Time Point | Statistic/<br>Category | Cohort 1<br>(n=XXX) | Cohort 2<br>(n=XXX) |
|---|---|---|---|---|---|
| All Subjects | Sitting Diastolic BP (mmHg) | Screening | N | XX | XX |
| | | | Mean (SD) | XX (XX.X) | XX (XX.X) |
| | | | Median | XX | XX |
| | | | Range | XX, XX | XX, XX |
| | | Day 0 Initial (Baseline) | N | XX | XX |
| | | | Mean (SD) | XX (XX.X) | XX (XX.X) |
| | | | Median | XX | XX |
| | | | Range | XX, XX | XX, XX |
| | | 72hr / Day 3 | N | XX | XX |
| | | | Mean (SD) | XX (XX.X) | XX (XX.X) |
| | | | Median | XX | XX |
| | | | Range | XX, XX | XX, XX |
| | | Change from Baseline at 72hr / Day 3 | N | XX | XX |
| | | A Substitute at 12m 1 2m 2 | Mean (SD) | XX (XX.X) | XX (XX.X) |
| | | | Median | XX | XX |
| | | | Range | XX, XX | XX, XX |
| | | Day 14 | N | XX | XX |
| | | 24, 11 | Mean (SD) | XX (XX.X) | XX (XX.X) |
| | | | Median | XX | XX |
| | | | Range | XX, XX | XX, XX |
| | | Change from Baseline at Day 14 | N | XX | XX |
| | | 8 | Mean (SD) | XX (XX.X) | XX (XX.X) |
| | | | Median | XX | XX |
| | | | Range | XX, XX | XX, XX |
| | | Day 28 | N | XX | XX |
| | | <b>,</b> | Mean (SD) | XX (XX.X) | XX (XX.X) |
| | | | Median | XX | XX |
| | | | Range | XX, XX | XX, XX |
| | | Change from Baseline at Day 28 | N | XX | XX |
| | | | Mean (SD) | XX (XX.X) | XX (XX.X) |
| | | | Median | XX | XX |
| | | | Range | XX, XX | XX, XX |
| | | Day 35 (End of Study) | N | XX | XX |
| | | , . , (, ) | Mean (SD) | XX (XX.X) | XX (XX.X) |
| | | | Median | XX | XX |
| | | | Range | XX, XX | XX, XX |
| | | Change from Baseline at Day 35 (End of Study) | N | XX | XX |
| | | and the state of t | Mean (SD) | XX (XX.X) | XX (XX.X) |
| | | | Median | XX | XX |
| | | | Range | XX, XX | XX, XX |


| Age Group Vital Sign | Time Point | Statistic/<br>Category | Cohort 1 (n=XXX) | Cohort 2<br>(n=XXX) |
|---|---|---|---|---|
| Note to programmer, repeat above for Systolic | BP, Heart Rate, and for two age stratu | m: 1 - < 6 years, and 6 - 17 years | . Note also that | height and |


# **Table of Contents**

| Listing 16.2.1.1 Completion/Discontinuation. |
|---|
| Listing 16.2.1.2 Identification of Subjects with Clinically Important Protocol Violations |
| Listing 16.2.1.3 Inclusion/Exclusion Criteria |
| Listing 16.2.1.4 Patient Populations |
| Listing 16.2.1.5 Demographics |
| Listing 16.2.1.6 Medical/Surgical History |
| Listing 16.2.1.7 Drug Allergy/Intolerance at Screening. |
| Listing 16.2.1.8 IV Iron Intolerance |
| Listing 16.2.1.9 Physical Examination |
| Listing 16.2.1.10 Iron Deficiency |
| Listing 16.2.2.1 Erythropoiesis Stimulating Agent |
| Listing 16.2.2.2 Ferric Carboxymaltose Administration |
| Listing 16.2.2.3 Pharmacokinetic Samples |
| Listing 16.2.3.1 Concomitant Medications |
| Listing 16.2.3.2.1 Central Laboratory Values - CFR |
| Listing 16.2.3.2.2 Central Laboratory Values – Lab Transfer |
| Listing 16.2.3.2.3 Potentially Clinically Significant Central Laboratory Values – Lab Transfer |
| Listing 16.2.3.3.1 Vital Signs |
| Listing 16.2.3.4 Adverse Event Details |


## Listing 16.2.1.1 Completion/Discontinuation

| ite/ | Safety | PK | Group | Date of<br>First<br>Dose | Date of Completion or Discontinuation (RxDay) | Subject<br>Status | Physician<br>Decision,<br>Specify | If<br>Other,<br>Specify | Date of<br>Death<br>(RxDay) | Autopsy | Primary<br>Cause of<br>Death | Pregnant<br>During<br>Study | Lactation<br>Exposure | Inter-<br>vention | Date | Increase in Dose of Erythrop- oletin for any Reason |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | | | | • | • | | | |
| - | | | | | | | | | | | | | -11 | | | |
| | | | | | | Listing 16.2 | 2.1.2 Identific | cation of Su | bjects with | Clinically In | nportant Pro | otocol Violat | ions | | | |
| | Site | / Subject | Safety | y Pk | C Group | Clinically In | portant Prote | ocol Violatio | n | | | | | | | |

## Listing 16.2.1.3 Inclusion/Exclusion Criteria

| te/ Subject | Safety | PK | Group | Did subject meet all inclusion and exclusion criteria? | Inclusion | /Exclusion Cat<br>Not Met | tegory | | Exclusion Numb | er Gr | /aiver<br>anted?<br>Y/N | Waiver Date | Waiver<br>Granted b |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | Listing 1 | 6.2.1.4 Patient | Popula | ations | <b>9</b> - | | | | |
| | | | | Site/ Subje | ect Group | Safety Popul | ation | PK/PD Pop | ulation_ | | | | |
| | | | | - | | | | | | | | | |
| | | | | | Listing | g 16.2.1.5 Dem | ograph | nics | | | | | |
| | | | | | | Age (yrs) | | Ethnicity<br>(Hispanic | American | | | Native | |
| Site/ Subjec | • 5- | ıfety | PK | Group B | irth Date | at Date of Screening | Sex | or<br>Latino) | Indian/Alaska<br>Native | Asian | Black/Afric | an Hawaiian/Ot | |


| Site/Subject Safety PK Group Body System Medical Condition/Past Surgery | Start Date | End Date | Ongoing? |
|---|---|---|---|
| Listing 16.2.1.7 Drug Allergy/Intoleran | nce at Screen | ning | |
| ite/ Subject Safety PK Group Does the subject have any drug allergies/intolerance | Drug/Drug | g Class Re | action Symptom |


## Listing 16.2.1.8 IV Iron Intolerance

| ite/ Subject | Safety | PK | Group | | | on intolerance? | If y | es, Name | Itching | g Rasl | n Br | onchospasm | Hypotensio | on C | )ther | Sodium Ferr<br>Other Symp | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | Listing 16.2. | 1.9 Physical 1 | Examinatio | n | | | | | | |
| | | | | Site/ S | Subject | Group Vis | it Exam Per | rformed? Bod | ly System ] | Not Done | Result | Specify Abnor | malities | | | | |
| | | | | - | | | | | | | | | | | | | |
| | | | | | | | | isting 16.2.1.10 | Iron Deficie | псу | | | | | | | |
| Site/ | | Group | Heavy<br>Uterine<br>Bleeding<br>Type | Polvps | Endo-<br>crine Dys-<br>function | Heavy<br>Uterine<br>Bleeding<br>Other | Heavy<br>Uterine<br>Bleeding<br>Specify | Gastro-<br>intestinal<br>Related<br>Symptom | Mal-<br>absorp-<br>tion | Celiac<br>Disease | GI<br>Bleed-<br>ing | Gastro-<br>intestinal<br>Other | Gastro-<br>intestinal<br>Specify | Cancer<br>Specify | Trauma<br>Specify | Surgery<br>Specify | Other<br>Specif |


## Listing 16.2.2.1 Erythropoiesis Stimulating Agent

| Site/<br>Subject | Safety P | PK Gr | oup | | Is subject using Er | ythropoiesis Sti | mulating A | Agent (ESA)? | | Has the c | lose been stable p<br>usion criteria? |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | Listing 16 | .2.2.2 Ferric C | arboxyma | ltose Administrat | on | | |
| ite/ Subject | Safety | PK | Group | Date | Total Dose Required for Injection | Start Time | Stop<br>Time | Total Dose of<br>Elemental Iron<br>Administered | IV<br>Administration | Reason Not<br>Administered | Other Specif |
| _ | | | | | | Listing 1 | 6.2.2.3 Pha | armacokinetic Sa | nples | | |
| | Site/<br>Subject | | Safety | PK | Group | | Timepoint | Not Done | Date (RxDay) | Time | |
| - | | | | | | | | | | | |
| - | | | | | | | | | | | |

-

#### Listing 16.2.3.1 Concomitant Medications

| Site/<br>Subject Safe | ety PK | Group | medications taken<br>from 30 days prior to<br>consent through end<br>of study or Day 35? | Drug<br>Name | Dose | Unit | Route | Other<br>Route | Indication | Start Date<br>(RxDay) | Stop Date<br>(RxDay) | Ongoing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|---|---|---|---|---|---|

## Listing 16.2.3.2.1 Central Laboratory Values - CFR


#### Listing 16.2.3.2.2 Central Laboratory Values - Lab Transfer

| | | Lis | sting 16.2.3 | .2.3 Potenti | ally Clinically Significant ( | Central Laboratory | Values – Lab T | ransfer | |
|---|---|---|---|---|---|---|---|---|---|
| Site/<br>Subject | Safety | PK | Group | Visit | Date (RxDay) | Lab | Result | Normal<br>Range | H/L<br>Flag |


## Listing 16.2.3.3.1 Vital Signs

| Site/ | | | | | | | | Not | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Site/<br>Subject | Safety | PK | Group | Visit | Vital Signs Collected? | Date (RxDay)/Time | Test | Done | Result | Units |
| doject | outery | 111 | Отобр | VIDIC | vitar organi comocioa. | Date (IdiDa) // Inite | 1000 | 20 | 1100011 | 01110 |

## Listing 16.2.3.4 Adverse Event Details

| | | | | | Onset | Resolution | | CTC | == | | | | | Did the AE result in the |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | Date | Date | | Toxicity | Action | | Other | | | subject being |
| Site/ | | | Any Verbatim | | (RxDay) | (RxDay)/ | | Criteria | Taken With | | Treatment, | Final | | discontinued form the |
| Subject Safety | PK | Group | AE? Term | Serious | / Time | Time | Continuing | Grade | Study Drug | Treatment | Specify | Outcome | Causality | study? |

